CLINICAL TRIAL: NCT06388967
Title: Early Detection of Pancreatic Cancer: Prospective Study
Brief Title: Pancreatic Cancer Detection Consortium
Acronym: PCDC
Status: Recruiting | Type: Observational
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 19288/PCDC
Record Dates: First submitted 2024-04-19; First posted 2024-04-29 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Pancreatic Cancer; Pancreatic Carcinoma; Pancreatic Adenocarcinoma; Pancreatic Ductal Adenocarcinoma; Pancreatic Neoplasms; Pancreatic Cancer Stage I; Pancreatic Cancer Stage; Pancreatic Cancer Resectable; Pancreatic Cancer Stage 0; Pancreatic Cancer Stage II; Pancreatic Cancer Stage III; Pancreatic Cancer, Adult; Pancreatic Cancer Non-resectable
Keywords: Micro RNA; Exosome; Cell free; Early detection; Screening
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatic cancer, adult

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Patients with Pancreatic Cancer Ductal Adenocarcinoma (Training): Individuals diagnosed with pancreatic ductal adenocarcinoma
  Interventions: Diagnostic Test: PANcreatic cancer Exosome Early detectiON (PANXEON)
- Individuals without Pancreatic Cancer Ductal Adenocarcinoma (Training): Individuals without pancreatic ductal adenocarcinoma
  Interventions: Diagnostic Test: PANcreatic cancer Exosome Early detectiON (PANXEON)
- Patients with Pancreatic Cancer Ductal Adenocarcinoma (Validation): Individuals diagnosed with pancreatic ductal adenocarcinoma
  Interventions: Diagnostic Test: PANcreatic cancer Exosome Early detectiON (PANXEON)
- Individuals without Pancreatic Cancer Ductal Adenocarcinoma (Validation): Individuals without pancreatic ductal adenocarcinoma
  Interventions: Diagnostic Test: PANcreatic cancer Exosome Early detectiON (PANXEON)

INTERVENTIONS:
Diagnostic Test: PANcreatic cancer Exosome Early detectiON (PANXEON) — This test will utilize quantitative reverse transcriptase polymerase chain reaction (qRT-PCR) to quantify the expression levels of 5 cell-free and 8 exosome-miRNAs in plasma samples obtained from patients with pancreatic ductal adenocarcinoma and from individuals without it
  Other Names: PANXEON (PANcreatic cancer Exosome Early detectiON)

SUMMARY:
This study aims to prospective validate an exosome-based miRNA signature for noninvasive and early detection of pancreatic ductal adenocarcinoma.

DETAILED DESCRIPTION:
Pancreatic ductal adenocarcinoma (PDAC) is one of the deadliest forms of cancer. It often goes undetected until it is at an advanced stage, making it challenging to treat. Currently, only a small percentage of patients are diagnosed early enough for effective treatment. While a blood marker exists, called serum carbohydrate antigen 19-9 (CA19-9), it is used primarily to track the disease, and it is unreliable for early detection.

To address this problem, the researchers have developed a new method to analyze circulating vesicles (called exosomes), which contain specific genetic material called microRNAs (miRNAs). In a previous study, by analyzing both the miRNAs that circulate freely in serum and the miRNAs that are inside the exosomes, the researchers have already identified a combination of 13 miRNAs that could accurately detect early-stage PDAC.

In this study, the researchers will test this method in a larger international cohort study. This study aims to confirm the effectiveness of this approach in identifying PDAC at its earliest stages.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of pancreatic ductal adenocarcinoma, stages I-IV (TNM classification, 8th edition)
* Received standard diagnostic and staging procedures as per local guidelines, and at least one sample was drawn before receiving any curative-intent treatment.
* Imaging- or endoscopy-based proof of lack of pancreatic ductal adenocarcinoma at the time of sampling (Non-disease controls)

Exclusion Criteria:

* Lack of written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Independent cohorts of individuals with and without pancreatic cancer (cases and controls, respectively)
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2026-06-18 (Estimated); Study Completion 2026-06-18 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | Through study completion, an average of 1 year
  True positive rate: the probability of a positive test result, conditioned on the individual truly being positive

SECONDARY OUTCOMES:
Specificity | Through study completion, an average of 1 year
  True negative rate: the probability of a negative test result, conditioned on the individual truly being negative
Accuracy | Through study completion, an average of 1 year
  A measure of trueness: proportion of correct predictions (both true positives and true negatives) among the total number of cases examined

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Goel, PhD, Principal Investigator — City of Hope Medical Center
Locations (11):
- United States (9):
  - Translational Genomics Research Institute, Phoenix, Arizona
  - Honorhealth, Scottsdale, Arizona
  - City of Hope Medical Center, Monrovia, California
  - Hoag Center, Newport Beach, California
  - OSF HealthCare, Peoria, Illinois
  - Ochsner Medical Center, Jefferson, Louisiana
  - Atlantic Health System, Morristown, New Jersey
  - Piedmont Medical Center, Rock Hill, South Carolina
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Nagoya University, Nagoya, Japan
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
Data collected for the study will be made available to others, including de-identified participant data, at publication, via a signed data access agreement and at the discretion of the investigators' approval of the proposed use of such data

REFERENCES:
- [Background] Ryan DP, Hong TS, Bardeesy N. Pancreatic adenocarcinoma. N Engl J Med. 2014 Sep 11;371(11):1039-49. doi: 10.1056/NEJMra1404198. No abstract available. PMID 25207767
- [Background] Kleeff J, Korc M, Apte M, La Vecchia C, Johnson CD, Biankin AV, Neale RE, Tempero M, Tuveson DA, Hruban RH, Neoptolemos JP. Pancreatic cancer. Nat Rev Dis Primers. 2016 Apr 21;2:16022. doi: 10.1038/nrdp.2016.22. PMID 27158978
- [Background] Mizrahi JD, Surana R, Valle JW, Shroff RT. Pancreatic cancer. Lancet. 2020 Jun 27;395(10242):2008-2020. doi: 10.1016/S0140-6736(20)30974-0. PMID 32593337
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Rahib L, Smith BD, Aizenberg R, Rosenzweig AB, Fleshman JM, Matrisian LM. Projecting cancer incidence and deaths to 2030: the unexpected burden of thyroid, liver, and pancreas cancers in the United States. Cancer Res. 2014 Jun 1;74(11):2913-21. doi: 10.1158/0008-5472.CAN-14-0155. PMID 24840647
- [Background] Vincent A, Herman J, Schulick R, Hruban RH, Goggins M. Pancreatic cancer. Lancet. 2011 Aug 13;378(9791):607-20. doi: 10.1016/S0140-6736(10)62307-0. Epub 2011 May 26. PMID 21620466
- [Background] Uesaka K, Boku N, Fukutomi A, Okamura Y, Konishi M, Matsumoto I, Kaneoka Y, Shimizu Y, Nakamori S, Sakamoto H, Morinaga S, Kainuma O, Imai K, Sata N, Hishinuma S, Ojima H, Yamaguchi R, Hirano S, Sudo T, Ohashi Y; JASPAC 01 Study Group. Adjuvant chemotherapy of S-1 versus gemcitabine for resected pancreatic cancer: a phase 3, open-label, randomised, non-inferiority trial (JASPAC 01). Lancet. 2016 Jul 16;388(10041):248-57. doi: 10.1016/S0140-6736(16)30583-9. Epub 2016 Jun 2. PMID 27265347
- [Background] Conroy T, Hammel P, Hebbar M, Ben Abdelghani M, Wei AC, Raoul JL, Chone L, Francois E, Artru P, Biagi JJ, Lecomte T, Assenat E, Faroux R, Ychou M, Volet J, Sauvanet A, Breysacher G, Di Fiore F, Cripps C, Kavan P, Texereau P, Bouhier-Leporrier K, Khemissa-Akouz F, Legoux JL, Juzyna B, Gourgou S, O'Callaghan CJ, Jouffroy-Zeller C, Rat P, Malka D, Castan F, Bachet JB; Canadian Cancer Trials Group and the Unicancer-GI-PRODIGE Group. FOLFIRINOX or Gemcitabine as Adjuvant Therapy for Pancreatic Cancer. N Engl J Med. 2018 Dec 20;379(25):2395-2406. doi: 10.1056/NEJMoa1809775. PMID 30575490
- [Background] Conroy T, Desseigne F, Ychou M, Bouche O, Guimbaud R, Becouarn Y, Adenis A, Raoul JL, Gourgou-Bourgade S, de la Fouchardiere C, Bennouna J, Bachet JB, Khemissa-Akouz F, Pere-Verge D, Delbaldo C, Assenat E, Chauffert B, Michel P, Montoto-Grillot C, Ducreux M; Groupe Tumeurs Digestives of Unicancer; PRODIGE Intergroup. FOLFIRINOX versus gemcitabine for metastatic pancreatic cancer. N Engl J Med. 2011 May 12;364(19):1817-25. doi: 10.1056/NEJMoa1011923. PMID 21561347
- [Background] Von Hoff DD, Ervin T, Arena FP, Chiorean EG, Infante J, Moore M, Seay T, Tjulandin SA, Ma WW, Saleh MN, Harris M, Reni M, Dowden S, Laheru D, Bahary N, Ramanathan RK, Tabernero J, Hidalgo M, Goldstein D, Van Cutsem E, Wei X, Iglesias J, Renschler MF. Increased survival in pancreatic cancer with nab-paclitaxel plus gemcitabine. N Engl J Med. 2013 Oct 31;369(18):1691-703. doi: 10.1056/NEJMoa1304369. Epub 2013 Oct 16. PMID 24131140
- [Background] Golan T, Hammel P, Reni M, Van Cutsem E, Macarulla T, Hall MJ, Park JO, Hochhauser D, Arnold D, Oh DY, Reinacher-Schick A, Tortora G, Algul H, O'Reilly EM, McGuinness D, Cui KY, Schlienger K, Locker GY, Kindler HL. Maintenance Olaparib for Germline BRCA-Mutated Metastatic Pancreatic Cancer. N Engl J Med. 2019 Jul 25;381(4):317-327. doi: 10.1056/NEJMoa1903387. Epub 2019 Jun 2. PMID 31157963
- [Background] Fahrmann JF, Schmidt CM, Mao X, Irajizad E, Loftus M, Zhang J, Patel N, Vykoukal J, Dennison JB, Long JP, Do KA, Zhang J, Chabot JA, Kluger MD, Kastrinos F, Brais L, Babic A, Jajoo K, Lee LS, Clancy TE, Ng K, Bullock A, Genkinger J, Yip-Schneider MT, Maitra A, Wolpin BM, Hanash S. Lead-Time Trajectory of CA19-9 as an Anchor Marker for Pancreatic Cancer Early Detection. Gastroenterology. 2021 Mar;160(4):1373-1383.e6. doi: 10.1053/j.gastro.2020.11.052. Epub 2020 Dec 14. PMID 33333055
- [Background] Majumder S, Taylor WR, Foote PH, Berger CK, Wu CW, Mahoney DW, Bamlet WR, Burger KN, Postier N, de la Fuente J, Doering KA, Lidgard GP, Allawi HT, Petersen GM, Chari ST, Ahlquist DA, Kisiel JB. High Detection Rates of Pancreatic Cancer Across Stages by Plasma Assay of Novel Methylated DNA Markers and CA19-9. Clin Cancer Res. 2021 May 1;27(9):2523-2532. doi: 10.1158/1078-0432.CCR-20-0235. Epub 2021 Feb 16. PMID 33593879
- [Background] Gui JC, Yan WL, Liu XD. CA19-9 and CA242 as tumor markers for the diagnosis of pancreatic cancer: a meta-analysis. Clin Exp Med. 2014 May;14(2):225-33. doi: 10.1007/s10238-013-0234-9. Epub 2013 Mar 3. PMID 23456571
- [Background] Tempero MA, Uchida E, Takasaki H, Burnett DA, Steplewski Z, Pour PM. Relationship of carbohydrate antigen 19-9 and Lewis antigens in pancreatic cancer. Cancer Res. 1987 Oct 15;47(20):5501-3. PMID 3308077
- [Background] Martin LK, Wei L, Trolli E, Bekaii-Saab T. Elevated baseline CA19-9 levels correlate with adverse prognosis in patients with early- or advanced-stage pancreas cancer. Med Oncol. 2012 Dec;29(5):3101-7. doi: 10.1007/s12032-012-0278-9. Epub 2012 Jun 24. PMID 22729400
- [Background] Luo G, Liu C, Guo M, Cheng H, Lu Y, Jin K, Liu L, Long J, Xu J, Lu R, Ni Q, Yu X. Potential Biomarkers in Lewis Negative Patients With Pancreatic Cancer. Ann Surg. 2017 Apr;265(4):800-805. doi: 10.1097/SLA.0000000000001741. PMID 28267695
- [Background] Cescon DW, Bratman SV, Chan SM, Siu LL. Circulating tumor DNA and liquid biopsy in oncology. Nat Cancer. 2020 Mar;1(3):276-290. doi: 10.1038/s43018-020-0043-5. Epub 2020 Mar 20. PMID 35122035
- [Background] Pantel K, Alix-Panabieres C. Liquid biopsy and minimal residual disease - latest advances and implications for cure. Nat Rev Clin Oncol. 2019 Jul;16(7):409-424. doi: 10.1038/s41571-019-0187-3. PMID 30796368
- [Background] Crowley E, Di Nicolantonio F, Loupakis F, Bardelli A. Liquid biopsy: monitoring cancer-genetics in the blood. Nat Rev Clin Oncol. 2013 Aug;10(8):472-84. doi: 10.1038/nrclinonc.2013.110. Epub 2013 Jul 9. PMID 23836314
- [Background] Kilgour E, Rothwell DG, Brady G, Dive C. Liquid Biopsy-Based Biomarkers of Treatment Response and Resistance. Cancer Cell. 2020 Apr 13;37(4):485-495. doi: 10.1016/j.ccell.2020.03.012. PMID 32289272
- [Background] Bloomston M, Frankel WL, Petrocca F, Volinia S, Alder H, Hagan JP, Liu CG, Bhatt D, Taccioli C, Croce CM. MicroRNA expression patterns to differentiate pancreatic adenocarcinoma from normal pancreas and chronic pancreatitis. JAMA. 2007 May 2;297(17):1901-8. doi: 10.1001/jama.297.17.1901. PMID 17473300
- [Background] Jin X, Chen Y, Chen H, Fei S, Chen D, Cai X, Liu L, Lin B, Su H, Zhao L, Su M, Pan H, Shen L, Xie D, Xie C. Evaluation of Tumor-Derived Exosomal miRNA as Potential Diagnostic Biomarkers for Early-Stage Non-Small Cell Lung Cancer Using Next-Generation Sequencing. Clin Cancer Res. 2017 Sep 1;23(17):5311-5319. doi: 10.1158/1078-0432.CCR-17-0577. Epub 2017 Jun 12. PMID 28606918
- [Background] Yu W, Hurley J, Roberts D, Chakrabortty SK, Enderle D, Noerholm M, Breakefield XO, Skog JK. Exosome-based liquid biopsies in cancer: opportunities and challenges. Ann Oncol. 2021 Apr;32(4):466-477. doi: 10.1016/j.annonc.2021.01.074. Epub 2021 Feb 4. PMID 33548389
- [Background] Krug AK, Enderle D, Karlovich C, Priewasser T, Bentink S, Spiel A, Brinkmann K, Emenegger J, Grimm DG, Castellanos-Rizaldos E, Goldman JW, Sequist LV, Soria JC, Camidge DR, Gadgeel SM, Wakelee HA, Raponi M, Noerholm M, Skog J. Improved EGFR mutation detection using combined exosomal RNA and circulating tumor DNA in NSCLC patient plasma. Ann Oncol. 2018 Mar 1;29(3):700-706. doi: 10.1093/annonc/mdx765. PMID 29216356
- [Background] San Lucas FA, Allenson K, Bernard V, Castillo J, Kim DU, Ellis K, Ehli EA, Davies GE, Petersen JL, Li D, Wolff R, Katz M, Varadhachary G, Wistuba I, Maitra A, Alvarez H. Minimally invasive genomic and transcriptomic profiling of visceral cancers by next-generation sequencing of circulating exosomes. Ann Oncol. 2016 Apr;27(4):635-41. doi: 10.1093/annonc/mdv604. Epub 2015 Dec 17. PMID 26681674
- [Background] Ingenito F, Roscigno G, Affinito A, Nuzzo S, Scognamiglio I, Quintavalle C, Condorelli G. The Role of Exo-miRNAs in Cancer: A Focus on Therapeutic and Diagnostic Applications. Int J Mol Sci. 2019 Sep 21;20(19):4687. doi: 10.3390/ijms20194687. PMID 31546654
- [Result] Toiyama Y, Okugawa Y, Fleshman J, Richard Boland C, Goel A. MicroRNAs as potential liquid biopsy biomarkers in colorectal cancer: A systematic review. Biochim Biophys Acta Rev Cancer. 2018 Dec;1870(2):274-282. doi: 10.1016/j.bbcan.2018.05.006. Epub 2018 May 29. PMID 29852194
- [Result] Shigeyasu K, Toden S, Zumwalt TJ, Okugawa Y, Goel A. Emerging Role of MicroRNAs as Liquid Biopsy Biomarkers in Gastrointestinal Cancers. Clin Cancer Res. 2017 May 15;23(10):2391-2399. doi: 10.1158/1078-0432.CCR-16-1676. Epub 2017 Jan 31. PMID 28143873
- [Result] Nishiwada S, Cui Y, Sho M, Jun E, Akahori T, Nakamura K, Sonohara F, Yamada S, Fujii T, Han IW, Tsai S, Kodera Y, Park JO, Von Hoff D, Kim SC, Li W, Goel A. Transcriptomic Profiling Identifies an Exosomal microRNA Signature for Predicting Recurrence Following Surgery in Patients With Pancreatic Ductal Adenocarcinoma. Ann Surg. 2022 Dec 1;276(6):e876-e885. doi: 10.1097/SLA.0000000000004993. Epub 2021 Jun 16. PMID 34132691
- [Result] Nakamura K, Zhu Z, Roy S, Jun E, Han H, Munoz RM, Nishiwada S, Sharma G, Cridebring D, Zenhausern F, Kim S, Roe DJ, Darabi S, Han IW, Evans DB, Yamada S, Demeure MJ, Becerra C, Celinski SA, Borazanci E, Tsai S, Kodera Y, Park JO, Bolton JS, Wang X, Kim SC, Von Hoff D, Goel A. An Exosome-based Transcriptomic Signature for Noninvasive, Early Detection of Patients With Pancreatic Ductal Adenocarcinoma: A Multicenter Cohort Study. Gastroenterology. 2022 Nov;163(5):1252-1266.e2. doi: 10.1053/j.gastro.2022.06.090. Epub 2022 Jul 16. PMID 35850192